CLINICAL TRIAL: NCT03241641
Title: Switching From Tenofovir Disoproxil Fumarate(TDF) to Tenofovir AlaFenamide(TAF) vs. Maintaining TDF Monotherapy in Chronic Hepatitis B Patients With Genotypic Resistance to Adefovir or Entecavir
Brief Title: Switching From TDF to TAF vs. Maintaining TDF in Chronic Hepatitis B With Resistance to Adefovir or Entecavir.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Young-Suk Lim (Other)
Collaborators: Samsung Medical Center (Other); Korea University Guro Hospital (Other); Konkuk University Medical Center (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor-Investigator, Young-Suk Lim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-320-4390
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintaining TAF monotherapy (Experimental): - Tenofovir AlaFenamide (Vemlidy) Tablet, 25mg, Daily Oral, 96 weeks
  Interventions: Drug: Tenofovir Alafenamide
- Switching from TDF to TAF (Active Comparator): * Tenofovir Disoproxil Fumarate (Viread) Tablet, 300mg, Daily Oral, 48 weeks
  * Tenofovir AlaFenamide (Vemlidy) Tablet, 25mg, Daily Oral, 48 weeks
  Interventions: Drug: Tenofovir Alafenamide; Drug: Tenofovir Disoproxil Fumarate

INTERVENTIONS:
Drug: Tenofovir Alafenamide — 25mg, Daily Oral
  Other Names: Vemlidy
Drug: Tenofovir Disoproxil Fumarate — 300mg, Daily Oral
  Other Names: Viread
  Arms: Switching from TDF to TAF

SUMMARY:
Treatment of CHB patients with genotypic resistance to NUCs has been problematic due to the lack of data from randomized trials. Recently, two randomized trials comparing the efficacy of TDF monotherapy versus TDF and ETV combination therapy in CHB patients with documented genotypic resistance to adefovir (ADV) or ETV demonstrated TDF monotherapy was not statistically different in viral suppression at week 48 of treatment.1,2 The extension study based on the above two trials merged study subjects from these trials with changing from TDF and ETV combination group to TDF monotherapy to evaluate long-term efficacy and safety of TDF monotherapy for multidrug-resistant patients. At the time of merging of 192 subjects, by intention-to-treat analysis, 66.3% of TDF group and 68.0% of TDF-ETV group had virological response as determined by serum HBV DNA <15 IU/mL. (in press) Three year long-term follow up study showed that the proportion of virologic suppression increased to 76.8% and 72.2% in TDF-TDF and TDF/TDF-ETV groups, respectively( P=0.46). (in press)

TAF, a novel prodrug of tenofovir was developed to have greater stability in plasma than TDF, thereby enabling more efficient delivery of the active metabolite to target cells at a substantially lower dose. The reduced systemic exposure of tenofovir offers the potential for an improved safety profile compared to TDF a benefit that demonstrated in a recent clinical trial in patients with HIV infection. In a recent double-blind randomized phase 3 noninferiority trial with 873 treatment naive patients who were positive for HBeAg, the proportion of patients receiving TAF who had HBV DNA <29 IU/mL at week 48 was 64%, which was non-inferior to the rate of 67% in patients receiving TDF (P=0.25).3 In the safety profile, TAF group had significantly smaller decrease in BMD than TDF group in the hip and spine, as well as significantly smaller increases in serum creatinine at week 48.3 For treatment naive HBeAg negative patients, a recent study with 425 subjects applied the same methodology and showed noninferiority in efficacy of TAF compared to TDF at week 48.4 Considering noninferiority in efficacy and superior bone and renal safety from TAF, TAF might be considered preferred choice of NUC instead of TDF. However, it is still unknown whether TAF would show similar efficacy and safety profile in patients with multidrug-resistant CHB.

DETAILED DESCRIPTION:
Study objectives The objective of this study is to evaluate whether efficacy, safety, and tolerability (including bone and renal outcomes) were non-inferior in patients switched to a tenofovir alafenamide (TAF), compared with patients who remained on tenofovir disoproxil fumarate (TDF).

Study procedures This is a randomized, active-controlled, open-label, multicenter study to evaluate safety and non-inferior efficacy of switching from TDF 300 mg QD to TAF 25 mg QD for 48 weeks in chronic hepatitis B patients who have genotypic resistance to Adefovir/Entecavir.

174 subjects who complete the previous IN-US-174-0202/0205 studies will be randomized in a 1:1 ratio (A:B) to receive either TAF 25 mg QD or TDF 300 mg QD Case group: approximately 87 subjects administered TAF 25 mg QD Control group: approximately 87 subjects administered TDF 300 mg QD

The primary analysis will occur at Week 48 with the primary efficacy endpoint being newly achievement and maintenance of virologic response (HBV DNA <60 IU/mL at Week 48).

The duration of maintaining both arms is 48 weeks. All subjects who complete 48 weeks of treatment are eligible for participation in the open label TAF 25 mg extension period for an additional 48 weeks (through Week 96)

ELIGIBILITY:
Inclusion Criteria:All of below

1. Patient must have the ability to understand and sign a written informed consent form; consent must be obtained prior to initiation of study procedures
2. Male or female, 20 to 80 years of age
3. Compensated liver disease (Child-Pugh score < 8)
4. HBsAg positive at least 6 months or more
5. HBeAg positive or negative
6. Confirmation of ETV resistance mutation (rt184, rtS202, or rtM250) at the enrollment of IN-US-174-0202 study, or ADV resistance mutation (rtA181V, rtA181T or rtN236T) at the enrollment of IN-US-174-0205 study
7. Completion of the week 240 visit in studies IN-US-174-0202 or 0205 study and maintained on TDF 300 mg QD
8. Patient is willing and able to comply with all study requirements

Exclusion Criteria: Any of below

1. Co-infection with HCV, HDV, HIV
2. Abusing alcohol (more than 40 g/day) or illicit drugs
3. Abnormal hematological and biochemical parameters, including:

1) serum bilirubin >3 mg/dL 2) prothrombin time (INR) >1.5 3) serum albumin <2.8 g/dL 4) ascites, encephalopathy or variceal hemorrhage 5) Child-Pugh score ≥8

4. Received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study

5. Medical condition that requires concurrent use of systemic corticosteroid or other immunosuppressive agent

6. Received solid organ or bone marrow transplant

7. Known hypersensitivity to study drugs, metabolites, or formulation excipients

8. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the patient unsuitable for the study or unable to comply with dosing requirements

9. Use of investigational agents within 3 months of screening, unless allowed by the Sponsor or Investigator

10. A history of hepatocellular carcinoma (HCC) within 5 years of screening

11. A history treated malignancy (other than HCC) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding three years

12. Participation in another investigational drug trial

13. Pregnant or breastfeeding or willing to be pregnant

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with virologic response | At week 48 of treatment
  The proportion of patients who achieve virologic response (serum HBV DNA concentrations below 60 IU/mL)

SECONDARY OUTCOMES:
Proportion of patients with virologic response | At week 96 of treatment
  The proportion of patients who achieve virologic response (serum HBV DNA concentrations below 60 IU/mL)
The proportion of patients with HBV DNA less than 15 IU/mL | At week 48, and 96 of treatment
  The proportion of patients with HBV DNA less than 15 IU/mL
The proportion of patients with normal ALT | At week 24, 48, 72 and 96 of treatment
  The proportion of patients with normal ALT
The proportion of patients with HBeAg loss or seroconversion | At week 24, 48, 72 and 96 of treatment
  The proportion of patients with HBeAg loss or seroconversion
The proportion of patients with HBsAg loss or seroconversion | At week 24, 48, 72 and 96 of treatment
  The proportion of patients with HBsAg loss or seroconversion
The incidence of virologic breakthrough | At week 48, and 96 of treatment
  Virologic breakthrough is defined as the increases in HBV DNA levels ≥1 log10IU/mL from nadir on two consecutive tests during continued treatment
The proportion of patients with resistance mutations to Entecavir or Adefovir or Tenofovir | At week 48, and 96 of treatment
  The proportion of patients with resistance mutations to Entecavir or Adefovir or Tenofovir
Percentage change from baseline in hip and spine bone mineral density (BMD) | At week 24, 48, 72 and 96 of treatment
  Percentage change from baseline in hip and spine bone mineral density (BMD)
Percentage change from baseline in urine beta2-microglobulin | At week 24, 48, 72 and 96 of treatment
  Percentage change from baseline in urine beta2-microglobulin
Percentage change from baseline in urine protein to creatinine ratio | At week 24, 48, 72 and 96 of treatment
  Percentage change from baseline in urine protein to creatinine ratio
Percentage change from baseline in urine albumin to creatinine ratio | At week 24, 48, 72 and 96 of treatment
  Percentage change from baseline in urine albumin to creatinine ratio
Percentage change from baseline in serum creatinine | At week 24, 48, 72 and 96 of treatment
  Percentage change from baseline in serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, M.D.,Ph D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chae HB, Kim JH, Kim JK, Yim HJ. Current status of liver diseases in Korea: hepatitis B. Korean J Hepatol. 2009 Dec;15 Suppl 6:S13-24. doi: 10.3350/kjhep.2009.15.S6.S13. PMID 20037275
- [Result] Kim SR, Kudo M, Hino O, Han KH, Chung YH, Lee HS; Organizing Committee of Japan-Korea Liver Symposium. Epidemiology of hepatocellular carcinoma in Japan and Korea. A review. Oncology. 2008;75 Suppl 1:13-6. doi: 10.1159/000173419. Epub 2008 Dec 17. PMID 19092267
- [Result] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Result] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Result] Iloeje UH, Yang HI, Su J, Jen CL, You SL, Chen CJ; Risk Evaluation of Viral Load Elevation and Associated Liver Disease/Cancer-In HBV (the REVEAL-HBV) Study Group. Predicting cirrhosis risk based on the level of circulating hepatitis B viral load. Gastroenterology. 2006 Mar;130(3):678-86. doi: 10.1053/j.gastro.2005.11.016. PMID 16530509
- [Result] Chang TT, Lai CL, Kew Yoon S, Lee SS, Coelho HS, Carrilho FJ, Poordad F, Halota W, Horsmans Y, Tsai N, Zhang H, Tenney DJ, Tamez R, Iloeje U. Entecavir treatment for up to 5 years in patients with hepatitis B e antigen-positive chronic hepatitis B. Hepatology. 2010 Feb;51(2):422-30. doi: 10.1002/hep.23327. PMID 20049753
- [Result] Snow-Lampart A, Chappell B, Curtis M, Zhu Y, Myrick F, Schawalder J, Kitrinos K, Svarovskaia ES, Miller MD, Sorbel J, Heathcote J, Marcellin P, Borroto-Esoda K. No resistance to tenofovir disoproxil fumarate detected after up to 144 weeks of therapy in patients monoinfected with chronic hepatitis B virus. Hepatology. 2011 Mar;53(3):763-73. doi: 10.1002/hep.24078. Epub 2010 Dec 22. PMID 21374657
- [Result] Zoulim F, Durantel D, Deny P. Management and prevention of drug resistance in chronic hepatitis B. Liver Int. 2009 Jan;29 Suppl 1:108-15. doi: 10.1111/j.1478-3231.2008.01939.x. PMID 19207973
- [Result] Bartholomeusz A, Locarnini SA. Antiviral drug resistance: clinical consequences and molecular aspects. Semin Liver Dis. 2006 May;26(2):162-70. doi: 10.1055/s-2006-939758. PMID 16673294
- [Result] Lim YS, Yoo BC, Byun KS, Kwon SY, Kim YJ, An J, Lee HC, Lee YS. Tenofovir monotherapy versus tenofovir and entecavir combination therapy in adefovir-resistant chronic hepatitis B patients with multiple drug failure: results of a randomised trial. Gut. 2016 Jun;65(6):1042-51. doi: 10.1136/gutjnl-2014-308435. Epub 2015 Mar 23. PMID 25800784
- [Result] Lim YS, Byun KS, Yoo BC, Kwon SY, Kim YJ, An J, Lee HC, Lee YS. Tenofovir monotherapy versus tenofovir and entecavir combination therapy in patients with entecavir-resistant chronic hepatitis B with multiple drug failure: results of a randomised trial. Gut. 2016 May;65(5):852-60. doi: 10.1136/gutjnl-2014-308353. Epub 2015 Jan 16. PMID 25596179
- [Result] Chan HL, Fung S, Seto WK, Chuang WL, Chen CY, Kim HJ, Hui AJ, Janssen HL, Chowdhury A, Tsang TY, Mehta R, Gane E, Flaherty JF, Massetto B, Gaggar A, Kitrinos KM, Lin L, Subramanian GM, McHutchison JG, Lim YS, Acharya SK, Agarwal K; GS-US-320-0110 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of HBeAg-positive chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):185-195. doi: 10.1016/S2468-1253(16)30024-3. Epub 2016 Sep 22. PMID 28404091
- [Result] Buti M, Gane E, Seto WK, Chan HL, Chuang WL, Stepanova T, Hui AJ, Lim YS, Mehta R, Janssen HL, Acharya SK, Flaherty JF, Massetto B, Cathcart AL, Kim K, Gaggar A, Subramanian GM, McHutchison JG, Pan CQ, Brunetto M, Izumi N, Marcellin P; GS-US-320-0108 Investigators. Tenofovir alafenamide versus tenofovir disoproxil fumarate for the treatment of patients with HBeAg-negative chronic hepatitis B virus infection: a randomised, double-blind, phase 3, non-inferiority trial. Lancet Gastroenterol Hepatol. 2016 Nov;1(3):196-206. doi: 10.1016/S2468-1253(16)30107-8. Epub 2016 Sep 22. PMID 28404092
- [Derived] Byun KS, Choi J, Kim JH, Lee YS, Lee HC, Kim YJ, Yoo BC, Kwon SY, Gwak GY, Lim YS. Tenofovir Alafenamide for Drug-Resistant Hepatitis B: A Randomized Trial for Switching From Tenofovir Disoproxil Fumarate. Clin Gastroenterol Hepatol. 2022 Feb;20(2):427-437.e5. doi: 10.1016/j.cgh.2021.04.045. Epub 2021 May 4. PMID 33962041